CLINICAL TRIAL: NCT04975243
Title: Clinical Evaluation to Assess the Safety and Efficacy of GentleMax Pro™/GentleMax Pro Plus™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMP20001
Record Dates: First submitted 2021-06-22; First posted 2021-07-23 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Unwanted Fine Facial Hair
Keywords: Laser Hair Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Unwanted Fine Facial Hair (Experimental): Up to three (3) treatments with GentleMax Pro/ GentleMax Pro Plus TM for Laser Hair Removal
  Interventions: Device: GentleMax Pro Plus 755nm and 1064nm laser system

INTERVENTIONS:
Device: GentleMax Pro Plus 755nm and 1064nm laser system — The GentleMax Pro Plus is a 755nm and 1064nm laser system. The GentleMax Pro PlusTM is indicated for stable long-term or permanent hair reduction using varying spot sizes and fluences.

SUMMARY:
This clinical study is intended to evaluate the safety and efficacy of the GentleMax Pro Plus™ laser system for its intended use of hair removal while using short pulse durations to improve the efficacy of achieving permanent reduction of fine facial hairs.

DETAILED DESCRIPTION:
Prospective, non-randomized, open label trial to evaluate the safety and efficacy of the GentleMax Pro Plus™ laser system for its intended use of hair removal with variable pulse durations and spot sizes.

Up to 30 subjects may be enrolled in this study at one (1) investigational site. Subjects having difficult to treat unwanted fine facial hairs having Fitzpatrick skin type (FST) I to VI are eligible for this study.

In order to have a diverse sample of study subjects, the following criteria was established to ensure a wide array of skin types and race and ethnicities for data analysis. At least 15 subjects must have FST III to V. The remaining subjects can include other FST, but must still have fine facial hairs where permanent hair reduction is difficult to achieve with 3 ms pulses.

Participants will receive four (4) laser hair removal treatment visits (with maximum interval of 10 weeks in between treatment visits) depending on the treatment area and three (3) follow up visits (1 month, 3 month, and 6 month after final treatment).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older
2. Willingness to provide signed, informed consent to participate in the study
3. Presence of unwanted hair of desired characteristics and treatment location to be evaluated in this study
4. Willingness to adhere to study treatment and follow-up schedule
5. Willingness to adhere to post-treatment care instructions
6. Willingness to allow photographs and/or video of treated areas, and to release their use for scientific/educational and/or promotional/marketing purposes
7. Willing to abstain from any other procedures, medications or topicals in the study treatment areas for the duration of the study which the investigator deems would interfere with the study

Exclusion Criteria:

1. Pregnant, planning pregnancy during the study, or breast feeding
2. Blonde, grey, or white hair in subjects seeking hair removal
3. Tattooed skin in the intended treatment area
4. Active suntan in the intended treatment area
5. History of active Herpes Virus Simplex (HSV) or similar condition in the intended treatment area unless treated with prophylactic medication
6. History of melanoma
7. History of vitiligo in the intended treatment area
8. History of keloid or hypertrophic scar formation
9. History of Melasma in the intended treatment area or per Investigator's discretion
10. Severe immunosuppression resulting from medications and/or a medical condition that could impair healing after treatment
11. Open wound or infection in the intended treatment area
12. History of light induced seizure disorders
13. The subject is not suitable, in the opinion of the Investigator, for participation in the study due to inability to adhere to the study requirements, medical, or other reasons that could compromise the study integrity or subject safety
14. Dermatologic and/or cosmetic procedures including use of medications, or topicals in the intended treatment area(s) during a timepoint prior to the study that the investigator deems the subject unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in hair removal/ hair clearance | 12 Months
  Improvement in hair removal/ hair clearance quantified by hair counts taken within a portion of the treatment area
Incidence, severity, and relatedness of adverse events | 12 Months
  Analysis of the incidence, severity, and relatedness of adverse events to study treatment.

SECONDARY OUTCOMES:
Laser Hair Removal improvement | 12 Months
  Overall level of improvement in laser hair removal as measured by Investigator using a 5-point Global Aesthetic Improvement Scale (IGAIS) (1= Very Much Improved, 5= Worse)
Subject satisfaction with treatment results | 12 Months
  Overall subject satisfaction with study treatments as measured using a 5- point Subject Satisfaction Scale (1= Not Satisfied, 5= Very Satisfied)
Subject satisfaction with treatment results | 12 Months
  Overall subject satisfaction with study treatments as measured using a 5- point Subject Global Aesthetic Improvement Scale (SGAIS) (1= Very Much Improved, 5= Worse)

OTHER OUTCOMES:
Subject Pain Assessment | 6 months
  Measurement of Subject Pain Assessment post-treatment for all subjects, using an 11-point Numerical Rating Scale (0=no pain, 10=extreme pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Candela Institute of Excellence, Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No